CLINICAL TRIAL: NCT00765024
Title: Efficacy and Safety of Ivermectin Versus Albendazole for Chronic Strongyloidiasis
Brief Title: Ivermectin Versus Albendazole for Chronic Strongyloidiasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Atlantic Laboratory Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TM001-2008
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Chronic Strongyloidiasis
Keywords: strongyloidiasis, ivermectin, albendazole
MeSH Terms: conditions — Strongyloidiasis | interventions — Ivermectin; Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Albendazole (Active Comparator): Albendazole for 7 days
  Interventions: Drug: Albendazole
- ivermectin (Experimental): ivermectin 200 mcg/kg single dose
  Interventions: Drug: Ivermectin
- ivermectin 2 doses (Experimental): ivermectin 200 mcg/kg two doses in 2 weeks
  Interventions: Drug: ivermectin

INTERVENTIONS:
Drug: Ivermectin — single dose of 200 mcg/kg
  Other Names: stromectal
  Arms: ivermectin
Drug: ivermectin — two single dose of 200mcg/kg in 2 weeks
  Other Names: stromectal
  Arms: ivermectin 2 doses
Drug: Albendazole — Albendazole 7 days
  Arms: Albendazole

SUMMARY:
A prospective controlled trial to compare the efficacy and safety of 7-day albendazole, single dose ivermectin, and 2-single dose ivermectin in 72 patients with chronic strongyloidiasis will be conducted at Siriraj Hospital, Bangkok, Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive strongyloides larva in the stool

Exclusion Criteria:

* Pregnancy
* Lactating women
* Known allergy to any study drug

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
cure rate | 1 year

SECONDARY OUTCOMES:
safety | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yupin Suputtamongkol, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Derived] Suputtamongkol Y, Premasathian N, Bhumimuang K, Waywa D, Nilganuwong S, Karuphong E, Anekthananon T, Wanachiwanawin D, Silpasakorn S. Efficacy and safety of single and double doses of ivermectin versus 7-day high dose albendazole for chronic strongyloidiasis. PLoS Negl Trop Dis. 2011 May 10;5(5):e1044. doi: 10.1371/journal.pntd.0001044. PMID 21572981